CLINICAL TRIAL: NCT06790940
Title: Construction of a Psoriasis and Psoriatic Arthritis Diagnostic Model Based on Multidimensional Nail Information
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 224-243
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis (PsO); Psoriatic Arthritis; Palmoplantar Pustulosis (PPP); Plaque Psoriasis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The samples collected are nail segments from all fingers of the participants. Specifically, the samples are 1-2 millimeter segments excised from the distal edge of the nail plate, which is located at the terminal part of the nail body and serves as the border connecting the nail bed to the fingertip.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with psoriasis
  Interventions: Other: No intervention
- Non-psoriasis subjects
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, no intervention will be implemented.

SUMMARY:
Psoriasis is a globally prevalent chronic relapsing skin disease, characterized by its long duration and tendency to relapse. In addition to skin symptoms, it can also affect nails and joints, leading to pathological features such as pitting, leukonychia, red lunula, or severe nail dystrophy. Some patients with psoriasis may develop psoriatic arthritis. Psoriatic arthritis (PsA) is a chronic relapsing musculoskeletal disease, characterized by psoriatic skin lesions accompanied by axial and peripheral joint damage, and often associated with characteristic manifestations of psoriatic nails. These nail changes typically indicate more severe disease and poorer prognosis. However, current diagnostic methods largely depend on the experience and professional knowledge of clinicians, which are subjective and uncertain. Moreover, histopathological examination is invasive and can cause additional pain and inconvenience to patients.

To develop an effective, convenient, and non-invasive early diagnostic tool for psoriasis, our research team has conducted in-depth studies in the field of psoriasis-related diagnosis and predictive models. We have successfully developed a predictive model for psoriatic arthritis, including six key predictive factors: history of joint swelling, history of arthritis, history of swelling and pain in fingers or toes, nail involvement, genital involvement, and a history of long-term local use of corticosteroids. Clinicians can effectively assess the risk of psoriatic arthritis by obtaining information about these six factors from patients. The paper "Early detection of psoriatic arthritis in patients with psoriasis: construction of a multifactorial prediction model" was published in Front. Immunol (DOI: 10.3389/fimmu.2024.1426127).

Raman spectroscopy is a rapid, non-invasive molecular vibration detection method that has shown great potential in medical diagnostics. Studies have shown that Raman spectroscopy can distinguish normal and abnormal tissues at the molecular level and has been proven feasible in nail testing. For psoriasis, a disease that causes significant nail changes, Raman spectroscopy offers unique advantages.

Based on this background, our project will conduct a prospective observational study on psoriasis and psoriatic arthritis using multidimensional nail data. We will integrate Raman spectroscopy data of nails and multidimensional clinical information and apply artificial intelligence algorithms to develop a new diagnostic tool for psoriasis and psoriatic arthritis. This tool aims to improve the accuracy and efficiency of diagnosis, providing strong support for the early detection and precise treatment of psoriasis and psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria for patients with psoriasis:

1. Previous or first-time diagnosis o psoriasis; if previously diagnosed, no restrictions on prior treatments;
2. Age ≥ 18 and ≤ 80 years, with no gender restrictions;
3. Consent to participate in this study and sign an informed consent form.

Inclusion criteria for non-psoriasis control subjects:

(1) Patients who visit for other non-psoriasis skin conditions such as eczema or acne, and are confirmed by dermatologists not to have psoriasis; (3) Age ≥ 18 and ≤ 80 years, with no gender restrictions; (4) Consent to participate in this study and sign an informed consent form.

-

Exclusion criteria for patients with psoriasis:

1. Those with unsuitable nail conditions for collection: patients with amputated fingers due to trauma or other reasons, and patients with any nail that is severely broken and cannot be effectively collected.
2. Patients with severe mental illness or cognitive impairment, lacking personal decision-making capacity, and unsuitable for participation in clinical research.
3. Patients with severe systemic diseases.
4. Patients with a history of malignant tumors, as well as those with primary or secondary immunodeficiency and hypersensitivity.
5. Patients whom the researchers deem unsuitable for participation in this study for other reasons.

Exclusion criteria for non-psoriasis subjects:

1. Those with unsuitable nail conditions for collection: patients with amputated fingers due to trauma or other reasons, and patients with any nail that is severely broken and cannot be effectively collected.
2. Patients with severe mental illness or cognitive impairment, lacking personal decision-making capacity, and unsuitable for participation in clinical research.
3. Patients with severe systemic diseases.
4. Patients with a history of malignant tumors, as well as those with primary or secondary immunodeficiency and hypersensitivity.
5. Patients whom the researchers deem unsuitable for participation in this study for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study plans to select and include 155 patients with psoriasis from those visiting the Department of Dermatology at Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, affiliated with Shanghai University of Traditional Chinese Medicine, as the experimental group. Additionally, 155 patients who visit for non-psoriasis skin conditions such as eczema or acne, and have been professionally diagnosed and confirmed by doctors not to have psoriasis, will be chosen as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Raman data | 1 day (The collected nail samples will be placed on aluminum-coated slides for Raman spectroscopic analysis, and the Raman peak data will be exported to form a txt file.)

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | The researcher conducted a Psoriasis Area and Severity Index (PASI) assessment on the psoriasis subjects on the 1 day of sample collection.
Body Surface Area (BSA) | The researcher conducted a Body Surface Area (BSA) assessment on the psoriasis subjects on the 1 day of sample collection.
Modified Nail Psoriasis Severity Index (mNAPSI) | The researcher conducted a Modified Nail Psoriasis Severity Index (mNAPSI) assessment on the psoriasis subjects on the 1 day of sample collection.
Classification of Psoriatic Arthritis (CASPAR) | The researcher conducted a Classification of Psoriatic Arthritis (CASPAR) assessment on the psoriasis subjects on the 1 day of sample collection.